CLINICAL TRIAL: NCT05177029
Title: Interventional, Randomized, Double-Blind, Sequential-Part, Placebo-Controlled, Single- and Multiple-Dose Study Investigating Safety, Tolerability, and Pharmacokinetic Properties of Lu AG06466 in Healthy Young Japanese and Caucasian Subjects
Brief Title: Safety and Tolerability Study of Lu AG06466 in Healthy Young Japanese and Caucasian Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated for strategic reasons.
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 19891A
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: Lu AG06466 or Placebo (Experimental): Participants will receive single dose of Lu AG06466 capsule or matching placebo orally on Day 1.
  Interventions: Drug: Lu AG06466; Drug: Placebo
- Part B: Lu AG06466 or Placebo (Experimental): Participants will receive starting dose of Lu AG06466 capsule or matching placebo orally once daily from Day 1 to Day 4 followed by Lu AG06466 capsule or matching placebo at a titrated treatment dose orally once daily from Day 5 until Day 8. Participants will then receive LuAG06466 capsule or matching placebo at a higher assigned dose orally once daily from Day 9 to Day 15.
  Interventions: Drug: Lu AG06466; Drug: Placebo

INTERVENTIONS:
Drug: Lu AG06466 — Lu AG06466 will be administered per schedule specified in the arm.
Drug: Placebo — Placebo matching to Lu AG06466 will be administered per schedule specified in the arm.

SUMMARY:
The main goal of this study is to evaluate the effect of Lu AG06466 on the body and what the body does to Lu AG06466 after single and multiple doses to healthy Japanese and Caucasian participants.

DETAILED DESCRIPTION:
This sequential study will be divided in two parts, Part A and Part B.

Part A will consist of 3 cohorts (Cohorts A1, A2, and A3) in which participants will be randomized to receive a single dose of Lu AG046466 or a matching placebo orally. After completing the safety review of data from Cohort A1, the study will proceed in Cohorts A2 and A3, with an increased dose of Lu AG046466 or matching placebo being administered to Japanese and Caucasian participants.

Part B dosing will only be initiated after completion of Part A. Part B will consist of 1 cohort (Cohort B1), to which multiple dose of Lu AG046466 or matching placebo will be administered after dose titration.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a BMI ≥18.5 and ≤25 kilograms (kg)/square meter (m^2) or ≤30 kg/m^2 for Japanese and Caucasian participants, respectively, and a body weight ≥50 kilograms (kg) at the screening visit and at the baseline visit.
* The participant is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, a neurological examination, vital signs, electrocardiograms (ECG), and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The participant has taken disallowed medication <1 week prior to the first dose of study drug or <5 half-lives of the disallowed medication as concomitant use prior to the screening visit.
* The participant has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, hematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.
* The participant has had a clinically significant illness <4 weeks prior to the first dose of study drug.
* The participant has received a SARS-CoV-2 (COVID-19) vaccination <30 days prior to the first dose of study drug.

Note: Other inclusion and exclusion criteria may apply.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants With Adverse Events | Baseline up to Day 12
Part B: Number of Participants With Adverse Events | Baseline up to Day 26
Part A: Area Under the Plasma Concentration-Time Curve of Lu AG06466 and Metabolite Lu AG06988 From Zero to Infinity (AUC0-inf) | 0 (pre-dose) up to 48 hours post-dose on Day 1 to Day 3
Part B: Area Under the Plasma Concentration-Time Curve of Lu AG06466 and Metabolite Lu AG06988 in a Dosing Interval (AUC0-τ) | 0 (pre-dose) up to 24 hours post-dose on Day 15
Part A: Maximum Observed Plasma Concentration (Cmax) of Lu AG06466 and Metabolite Lu AG06988 | 0 (pre-dose) up to 48 hours post-dose on Day 1 to Day 3
Part B: Cmax of Lu AG06466 and Metabolite Lu AG06988 | 0 (pre-dose) up to 24 hours post-dose on Day 1 and Day 15
Part A: Nominal Time Corresponding to the Occurrence of Cmax (Tmax) of Lu AG06466 and Metabolite Lu AG06988 | 0 (pre-dose) up to 48 hours post-dose on Day 1 to Day 3
Part B: Tmax of Lu AG06466 and Metabolite Lu AG06988 | 0 (pre-dose) up to 24 hours post-dose on Day 1 and Day 15
Part A: Apparent Elimination Half-Life (t1/2) of Lu AG06466 and Metabolite Lu AG06988 | 0 (pre-dose) up to 48 hours post-dose on Day 1 to Day 3
Part B: t1/2 of Lu AG06466 and Metabolite Lu AG06988 | 0 (pre-dose) up to 48 hours post-dose on Day 1 to Day 17
Part A: Metabolic Ratio of AUC0-inf (MRAUC0-inf): AUC0-inf, Lu AG06988/AUC0-inf, Lu AG06466 | 0 (pre-dose) up to 48 hours post-dose on Day 1 to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (1):
- P-One Clinic, Keikokai Medical Corporation, Yokamachi Hachioji City, Tokyo, Japan